CLINICAL TRIAL: NCT03511989
Title: Transverse Maxillary Expansion With a Segmental Le Fort I Osteotomy or Surgically Assisted Rapid Maxillary Expansion (SARME)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Tue Lindberg Blæhr, Consultant Oral and Maxillofacial Surgery, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-20160057
Record Dates: First submitted 2017-10-26; First posted 2018-04-30 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Maxilla; Hypoplasia
MeSH Terms: conditions — Retrognathia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Bone Borne distractor (Active Comparator): The device being investigated, Boneborne distraction appliance
  Interventions: Device: Bone borne distractor
- Tooth borne distractor (Other): The control device Toothborne distraction appliance
  Interventions: Device: Tooth borne distractor
- Segmental LF1 osteotomy group 1 (No Intervention): Control Group, no stabilization of palatal vault
- Segmental LF1 osteotomy group 2 (Active Comparator): Testgroup, biodegradable plate at osteotomy site in palate
  Interventions: Procedure: Segmental LF1 Osteotomy group 1; Procedure: Segmental LF1 Osteotomy group 3
- Segmental LF1 osteotomy group 3 (Active Comparator): Testgroup, autologous bonegraft at palatal osteotomy site
  Interventions: Procedure: Segmental LF1 Osteotomy group 1; Procedure: Segmental LF1 Osteotomy group 2

INTERVENTIONS:
Device: Bone borne distractor — Bone borne distraction device
  Arms: Bone Borne distractor
Device: Tooth borne distractor — Tooth borne distraction device
  Arms: Tooth borne distractor
Procedure: Segmental LF1 Osteotomy group 1
  Arms: Segmental LF1 osteotomy group 2; Segmental LF1 osteotomy group 3
Procedure: Segmental LF1 Osteotomy group 2
  Arms: Segmental LF1 osteotomy group 3
Procedure: Segmental LF1 Osteotomy group 3
  Arms: Segmental LF1 osteotomy group 2

SUMMARY:
To assess transverse dental and skeletal expansion and stability after SLFIO with no fixation of the palatal vault compared to stabilization of the palatal vault with an autogenous bone block graft or fixation of the palatal osteotomy site with a biodegradable plate.

To assess transverse maxillary dental and skeletal expansion and stability after SARME with a TB distraction appliance compared to a BB distraction appliance.

DETAILED DESCRIPTION:
Background: Surgical correction of transverse maxillary hypoplasia, in adolescents and adults is considered the least stable orthognathic procedure. Different surgical techniques have been advocated to improve the transverse stability. However, the pattern of transverse dental and skeletal expansion and long-term stability after segmental Le Fort I osteotomy (SLFIO) and surgically assisted rapid maxillary expansion (SARME) have never been compared systematically with different fixation techniques or distraction appliances.

Purpose: Test the H0-hypothesis of no difference in transverse stability after SLFIO without fixation of the palatal vault compared to stabilizing with either a bone block graft or a biodegradable plate. Moreover, test the H0-hypothesis of no difference in transverse maxillary dental and skeletal expansion and stability after SARME with either a tooth-borne (TB) or a bone-borne (BB) distraction appliance.

Method: 60 patients scheduled for SLFIO are included in a randomized clinical trial and allocated into 3 groups; I) stabilization of the palatal vault with a bone block graft, II) fixation of the palatal vault with a biodegradable plate and III) no fixation of the palatal vault. Moreover, 30 patients undergoing SARME are randomly allocated to either a TB or a BB distraction appliance. Transverse expansion and stability is assessed by clinical and radiographic measurements evaluating differences between dental and skeletal expansion, the pattern of skeletal expansion and the long-term stability.

Primary impact goal: Long-term transverse maxillary stability after SLFIO and SARME.

ELIGIBILITY:
Inclusion Criteria:

Mature non-syndromic patients scheduled for transverse expansion of the maxilla

Exclusion Criteria:

Previous orthognathic surgery involving the maxilla Congenital maxillofacial deformities

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Skeletal relapse | 2 years
  Relapse in milimeters

SECONDARY OUTCOMES:
Dental relapse | 2 years
  Relapse in milimeters

CONTACTS AND LOCATIONS:
Overall Officials: Tue Blæhr, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No